CLINICAL TRIAL: NCT01345604
Title: Reducing Posterior Knee Pain Following Total Knee Arthroplasty Using an Intraoperative Posterior Cruciate Ligament (Transcruciate) Injection
Brief Title: Intraoperative Posterior Cruciate Ligament (Transcruciate) Injection After Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatoon Health Region (Other)
Responsible Party: Principal Investigator, Jacelyn Larson, Faculty, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCL block
Record Dates: First submitted 2011-04-28; First posted 2011-05-02 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Arthroplasty, Replacement, Knee
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Placebo Comparator)
  Interventions: Procedure: transcruciate injection of 20cc of normal saline
- Ropivicaine (Active Comparator)
  Interventions: Procedure: transcruciate injection of 20 cc of 0.5% Ropivacaine

INTERVENTIONS:
Procedure: transcruciate injection of 20cc of normal saline — Group 2 (control group) will receive a transcruciate injection of 20cc of normal saline through the posterior cruciate ligament during the procedure (in addition to a subarachnoid block and femoral nerve block pre-operatively).
  Arms: Saline
Procedure: transcruciate injection of 20 cc of 0.5% Ropivacaine — Group 1 (study group) will receive a transcruciate injection of 20 cc of 0.5% Ropivacaine through the posterior cruciate ligament during the procedure (in addition to a subarachnoid block and femoral nerve block pre-operatively).
  Arms: Ropivicaine

SUMMARY:
his study is being done because total knee replacements can leave patients with considerable pain after surgery. Therefore, many studies have been done to find the best ways to control knee pain after the surgery. Currently, a popular approach is to use many different techniques to control the pain. This includes injecting freezing (local anesthetic) into the spinal column (spinal anesthetic), injecting freezing close to the nerves of the knee and using various kinds of medications (e.g. narcotics and anti-inflammatory medications). Studies have shown using this a combination of techniques can reduce pain and allow earlier discharge from the hospital. However, one downside to this approach is it does not usually control the pain in the back of the knee. One new technique has been used to try and overcome this. This technique is called a "posterior cruciate ligament block" or "PCL block". It involves injecting a drug into the back of the knee which will block the nerves in this area. Sometimes the investigators refer to this as "freezing".

The purpose of our study is to determine whether this "PCL Block" will improve pain after the total knee replacement surgery. The investigators will also determine whether this technique will improve movement in the knee and lessen narcotic usage after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists' (ASA) physical status classification (ASA) I and II patients undergoing unilateral total knee arthroplasty at Saskatoon City Hospital
* Patients recruited from the practice of 4 orthopedic surgeons

Exclusion Criteria:

* Inability to obtain informed consent
* Simultaneous bilateral total knee arthroplasty or revision cases
* Preexisting neurological deficits in the distribution of the femoral nerve or known diagnosis of peripheral neuropathy
* Coagulopathies
* Infection either systemically or at the needle insertion sites
* Allergies to local anesthetics or opioids
* Patients with a history of narcotic dependency or chronic pain
* ASA III and IV
* Body Mass Index (BMI) > 40

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Knee flexion | up to one week postoperative

SECONDARY OUTCOMES:
Postoperative pain score | in PACU , on ward (baseline), and post-op day 1 & 2 at 10am & 6pm
  Pain scores will be recorded at rest and on attempt of achieving a 90 degree passive flexion of the knee.
Total narcotic consumption | up to 1 week postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Saskatoon City Hospital, Saskatoon, Saskatchewan, Canada